CLINICAL TRIAL: NCT03372746
Title: Generation of Induced Pluripotent Stem (iPS) Cell Lines From Skin Fibroblast Cells of Participants With Age-Related Macular Degeneration: An Ancillary Study to the Age-Related Eye Disease Study-2 (AREDS2)
Brief Title: Generation of Induced Pluripotent Stem (iPS) Cell Lines From Skin Fibroblast Cells of Participants With Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180027; 18-EI-0027
Record Dates: First submitted 2017-12-13; First posted 2017-12-14 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: AMD
Keywords: Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Participants across multiple sites with AMD from the original cohort of study participants enrolled in the AREDS2

SUMMARY:
Background:

Age-related macular degeneration (AMD) is the leading cause of blindness in the United States. Currently, there is no safe way to obtain cells from the eye to study. But researchers now can turn other types of cells, like skin or blood, into induced pluripotent stem (iPS) cells. These can be grown in a lab and turned into other types of cells, like cells from the eye. This will allow researchers to understand and treat diseases of the eye such as AMD.

Objectives:

To establish a bank of samples that can be changed into other cell types, such as eye cells, to better understand diseases such as AMD. Also to test drugs in order to treat various eye diseases.

Eligibility:

People who provided DNA samples in another protocol (07-EI-0025)

Design:

Participants will be screened with their data from the previous protocol. Participants with select genetic variants will be chosen and contacted via phone.

Participants will have a punch skin biopsy. The skin will be washed. A numbing medication will be injected. A small piece of skin will be removed with a biopsy tool. The site will be covered with a dressing. They will receive instructions on how to care for the area. They will have follow-up visits if needed for clinical care for the area.

Participants may be asked to return if their first sample did not provide enough cells for the lab.

Participants sample will be developed into eye cells. The cells will be used to understand diseases and test new drugs.

DETAILED DESCRIPTION:
Objective: This ancillary study will establish a repository of biospecimens to generate induced pluripotent stem (iPS) cells that can be differentiated into ocular cell types, to be used for study of molecular mechanisms of and development of treatments for age-related macular degeneration (AMD). This repository will allow the cells to be used to perform high throughput drug screens to identify novel potential therapeutic compounds. Although research involving multiple different ocular cell types from these patients may be performed, the vast majority of the work will be centered on the retinal pigment epithelium (RPE) and neural retina. RPE and/or neural retinal cells generated from the iPS cells of participants with AMD will be used to analyze molecular mechanisms involved in disease initiation and progression.

Study Population: We plan to recruit 100 participants across multiple sites with AMD from the original cohort of study participants enrolled in the AREDS2 who are returning for a 10 year in-clinic study visit and have donated DNA in the AREDS2 study. Up to two participants will be enrolled at NEI. Participants with the highest genetic burden as well as those with rare variants will be included in the population.

Design: A 520 blood sample will be collected from 350 participants with specific genetic variants that are identified prior to the start of the study. Up to 60 participants will be enrolled at NEI. All of these participants were previously enrolled in the AREDS2 protocol (07-EI-0025) and they are returning for a 10-year in-clinic study visit for further phenotyping and for assessing the long-term effects of the ARESD2 supplements. Collected samples will be used to analyze molecular mechanisms involved in disease initiation and progression. In addition, the iPS cell-derived ocular cells may be used to perform high throughput (HTP) drug screens aimed at suppressing the molecular phenotypes of the disease and to identify potential therapeutic agents for these diseases. This study will typically require only one visit by each participant.

Outcome Measures: The primary outcome is to develop a repository for iPS cells for investigators involved in vision research. Secondary outcomes include the assessment of potential therapies for the treatment of age related macular disorder (AMD). There are no specific participant-based clinical outcomes for this protocol. Participants will, in general, be seen only once for this protocol, as this is an ancillary study to the main study.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. AREDS2 participants who have provided DNA samples. A list will be generated based upon the results, picking the top GWAS results from this cohort.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant is able to provide 20 ml blood sample.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Participant is unable to comply with study procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 participants across multiple sites with AMD from the original cohort of study participants will be enrolled in the AREDS2 who are returning for a 10 year in-clinic study visit and have donated DNA in the AREDS2 study
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to develop a repository for iPS cells for investigators involved in vision research. | Ongoing

SECONDARY OUTCOMES:
Secondary outcomes include the assessment of potential therapies for the treatment of age related macular disorder (AMD). | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (14):
- United States (14):
  - Retina-Vitreous Associates Med Group, Beverly Hills, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Emory University Eye Center, Atlanta, Georgia
  - Retina Vitreous Associates of Kentucky, Lexington, Kentucky
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Elman Retina Group, P.A., Rosedale, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Vision Research ROPARD Foundation/Associated Retinal Consultants, Grand Rapids, Grand Rapids, Michigan
  - Vision Research ROPARD Foundation/Associated Retinal Consultants, Novi, Novi, Michigan
  - Charlotte Eye Ear Nose & Throat Associates, Charlotte, North Carolina
  - Casey Eye Institute, Portland, Oregon
  - Texas Retina Associates, Dallas, Texas
  - John Moran Eye Center, University of Utah, Salt Lake City, Utah
  - University of Wisconsin-Madison, Madison, Wisconsin